CLINICAL TRIAL: NCT01598233
Title: Effects of Intragastric Balloon on Bone, Metabolic and Respiratory Parameters
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Miguel Madeira, Principal investigator, Universidade Federal do Rio de Janeiro
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3056-CEP/HUPE
Record Dates: First submitted 2012-05-04; First posted 2012-05-15 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Overweight; Obesity; Metabolic Syndrome
MeSH Terms: conditions — Overweight; Obesity; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intragastric balloon (Experimental): Patients submitted to six-month intragastric balloon
  Interventions: Device: Silimed Intragastric balloon

INTERVENTIONS:
Device: Silimed Intragastric balloon — Intragastric balloon inflated with 650 ml of NaCl 0.9% mixed with 20 ml of methylene blue solution

SUMMARY:
The purpose of this study is to evaluate the effects of intragastric balloon on bone, metabolic and respiratory parameters in 50 patients with metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* metabolic syndrome (IDF criteria)

Exclusion Criteria:

* menopause
* older than 50 years
* diabetes mellitus

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2011-03; Primary Completion 2012-01 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Change in bone mineral density and body composition | Baseline and 6 months
  Bone mineral density and body composition by dual-energy X-ray absorptiometry (DXA)
Change in fasting and postprandial glucose | Baseline and 6 months
Change in Pulmonary function tests | Baseline and 6 months
  Pulmonary function tests consiste of spirometry, body plethysmograph, diffusing capacity for carbon monoxide (DLco), and respiratory muscle strength. Measurements are conducted using the Collins Plus Pulmonary Function Testing Systems (Warren E. Collins, Inc., Braintree, MA, USA).
Change in bone microarchitecture | Baseline and 6 months
  Bone microarchitecture by high-resolution peripheral quantitative computed tomography
Change in lipid profile | Baseline and 6 months
  Total cholesterol, triglycerides, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol, very low-density lipoprotein cholesterol

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Estadual do Rio de Janeiro, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] Guedes EP, Madeira E, Mafort TT, Madeira M, Moreira RO, de Mendonca LMC, de Godoy-Matos AF, Lopes AJ, Farias MLF. Impact of 6 months of treatment with intragastric balloon on body fat and quality of life in obese individuals with metabolic syndrome. Health Qual Life Outcomes. 2017 Oct 24;15(1):211. doi: 10.1186/s12955-017-0790-x. PMID 29065923
- [Derived] Guedes EP, Madeira E, Mafort TT, Madeira M, Moreira RO, Mendonca LM, Godoy-Matos AF, Lopes AJ, Farias ML. Impact of a 6-month treatment with intragastric balloon on body composition and psychopathological profile in obese individuals with metabolic syndrome. Diabetol Metab Syndr. 2016 Dec 19;8:81. doi: 10.1186/s13098-016-0197-6. eCollection 2016. PMID 28031749